CLINICAL TRIAL: NCT04498494
Title: Role of Electrocardiograms in Risk Stratification and Analysis of the Characteristics of ST Elevation in Acute Myocarditis: A Two-center Study
Brief Title: The Role of Electrocardiograms in Risk Stratification and Analysis of the Characteristics of ST Elevation in Acute Myocarditis: a 2-centre Study
Status: Completed | Type: Observational
Sponsor: Yuanli Lei (Other)
Responsible Party: Sponsor-Investigator, Yuanli Lei, principal Investigator, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: Yuanli2020
Record Dates: First submitted 2020-07-25; First posted 2020-08-04 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Myocarditis
MeSH Terms: conditions — Myocarditis | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- myocarditis: The diagnosis of acute myocarditis was confirmed by a recent history of gastrointestinal/upper respiratory tract infection and/or complaints of cardiac symptoms and increasing cardiac markers and/or presentation with a new abnormality of the 12-lead ECGcombined with at least one of the following: ⅰ) Active or borderline biopsy according to the Dallas criteria (13); ⅱ) positive infectious origin of ventricular dysfunction; ⅲ) delayed enhancement on cardiac MRI consistent with myocarditis; or ⅳ) serological tests, ECGs, ultrasonic cardiogram (UCG), coronary angiography and ventriculography to exclude acute myocardial infarction (AMI), stress cardiomyopathy, congenital heart disease, myocarditis secondary to sepsis, valve disease, hyperthyroidism, autoimmune disease and rheumatic fever
  Interventions: Device: ECG
- fulminant myocarditis: In patients with acute myocarditis, a diagnosis of FM was determined upon identification of one or more of the following: Haemodynamic instability due to cardiogenic shock or arrhythmia; left ventricular dysfunction and low cardiac output syndrome requiring inotropes or mechanical circulatory support; mechanical ventilation; and/or cardiac arrest (CA)
  Interventions: Device: ECG

INTERVENTIONS:
Device: ECG — 12-lead ECG

SUMMARY:
The purpose of the present study was to investigate ECG findings of patients with acute myocarditis, ECG findings associated with fulminant myocarditis, and the characteristics of ST-elevation on admission.

DETAILED DESCRIPTION:
Acute myocarditis is a severe disease with high mortality rate and various dynamic changes visible on electrocardiograms (ECGs). The aim were to investigate ECG findings in acute myocarditis, ECG findings associated with fulminant myocarditis (FM), and the characteristics of ST elevation at admission. A retrospective analysis of 1814 ECGs was conducted from 274 consecutive patients with acute myocarditis aged ≥13 years, who were hospitalized in two centres between August 2007 and November 2019. All ECG obtained during the hospital course were evaluated by 2 electrophysiologists. A chi-square test was used to evaluate and compare the abnormal ECG findings between the FM and non-FM groups, and multivariate logistic regression analysis was performed to further evaluate ECG findings associated with FM. The Mann-Whitney U test was used to compare the duration of cardiac symptoms before admission for ST elevation at admission.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Acute myocarditis

  * complete data of ECG

Exclusion Criteria :

* Incomplete data;

  * a history of congenital heart disease, cardiomyopathy or arrhythmias;

    * myocarditis not being the primary diagnosis for a particular admission;

      * absence of cardiac symptoms.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 20 million residents of the South of Zhejiang Province
Sampling Method: Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
The percentage rate of ST elevation | through study completion, an average of 2 years
  ST elevation was the typical ECG changes of acute myocarditis. The study was to investigate how many patients presented with ST elevation on admission.

SECONDARY OUTCOMES:
Atrioventricular block, ventricular tachycardia and their correlationwith Fulminant myocarditis (FM) | through study completion, an average of 6 months
  FM is a peculiar clinical condition and is an acute and severe form of myocarditis . FM is associated with a wide variety of ECG findings. The study was to investigate Atrioventricular block, ventricular tachycardia and their correlation with FM.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] JCS Joint Working Group. Guidelines for diagnosis and treatment of myocarditis (JCS 2009): digest version. Circ J. 2011;75(3):734-43. doi: 10.1253/circj.cj-88-0008. Epub 2011 Feb 4. No abstract available. PMID 21304213
- [Background] Caforio AL, Pankuweit S, Arbustini E, Basso C, Gimeno-Blanes J, Felix SB, Fu M, Helio T, Heymans S, Jahns R, Klingel K, Linhart A, Maisch B, McKenna W, Mogensen J, Pinto YM, Ristic A, Schultheiss HP, Seggewiss H, Tavazzi L, Thiene G, Yilmaz A, Charron P, Elliott PM; European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Current state of knowledge on aetiology, diagnosis, management, and therapy of myocarditis: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 Sep;34(33):2636-48, 2648a-2648d. doi: 10.1093/eurheartj/eht210. Epub 2013 Jul 3. PMID 23824828